CLINICAL TRIAL: NCT04573296
Title: Impact of Digital Therapeutic Intervention on Metabolic Parameters in Obese Adults With Insulin Resistance, Prediabetes and Type 2 Diabetes as Compared to Conventional Intensive Obesity Management Programme
Brief Title: Impact of Digital Therapeutic on Metabolic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitadio s.r.o. (Industry)
Collaborators: University Hospital Olomouc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Insulin Resistance; Prediabetic State; Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Insulin Resistance; Prediabetic State; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: This prospective randomized controlled study evaluates efficacy of lifestyle intervention using digital application Vitadio as compared to conventional high-intensity lifestyle intervention program administered at a specialized clinic at a University hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants using Vitadio (Experimental): Participants in the intervention arm undergo a 6-month digitally administered behavioral change program Vitadio focused on lifestyle change and self-management. The program aims for strengthening patients autonomy with the goal to promote weight loss and improve metabolic health. The program includes personalized education, adaptive daily tasks and weekly goals, automated motivational and educational messaging, monitoring tools, recipes, peer-support group and one-on-one remote coaching. In addition, they undergo regular face-to-face medical assessment.
  Interventions: Device: Vitadio
- Participants assigned to conventional high-intensity lifestyle intervention program (Active Comparator): Participants in the control group undergo a 6-month high-intensity lifestyle intervention program consisting of of 5 face-to-face nutrition/lifestyle education sessions. Participants can use an online diary tool for recording meals with an option to receive remote feedback on their diet from the educator. In addition, they undergo regular face-to-face medical assessment.
  Interventions: Behavioral: Conventional high-intensity lifestyle intervention program

INTERVENTIONS:
Device: Vitadio — A 6-month digitally administered behavioral change program Vitadio focus on lifestyle change and self-management. The program aims for strengthening patients autonomy with the goal to promote weight loss and improve metabolic health. The program includes personalized education, adaptive daily tasks and weekly goals, automated motivational and educational messaging, monitoring tools, recipes, peer-support group and remote coaching.
  Arms: Participants using Vitadio
Behavioral: Conventional high-intensity lifestyle intervention program — A 6-month high-intensity lifestyle intervention program consisting of 5 face-to-face nutrition/lifestyle education sessions. Participants can use an online diary tool for recording meals with an option to receive remote feedback on their diet from the educator.
  Arms: Participants assigned to conventional high-intensity lifestyle intervention program

SUMMARY:
The purpose of this prospective randomized controlled study is to evaluate the impact of a six-month digitally administered behavioral change program on body weight, glycemic control and other metabolic parameters in obese adults with insulin resistance, prediabetes or type 2 diabetes as compared to conventional high-intensity lifestyle intervention program administered at a specialized department of a university hospital.

DETAILED DESCRIPTION:
In this prospective randomized clinical study, obese adults with insulin resistance, prediabetes or diabetes mellitus type 2, patients of the Department of Exercise Medicine and Cardiovascular Rehabilitation at the University Hospital Olomouc, are randomized to receive either Vitadio or a conventional 6-month high-intensity lifestyle intervention program at the clinic.

Vitadio is a mobile application delivering behavioral change program focused on lifestyle change and self-management. The program aims for strengthening patients autonomy with the goal to promote weight loss and improve metabolic health. The program includes personalized education, adaptive daily tasks and weekly goals, automated motivational and educational messaging, monitoring tools, recipes, peer-support group and one-on-one remote coaching. Personalization of the intervention is achieved by analyzing participant's interactions with the application.

The conventional therapy consists of 5 face-to-face nutrition/lifestyle education sessions (at baseline, at 1st, 2nd and 3rd month, and at month 6). Participants in the control group can use an online diary tool for recording meals with an option to receive remote feedback on their diet from the educator. In addition, all participants undergo a regular medical assessment at the clinic (baseline, month 3, month 6).

The aim of the study is to assess feasibility and efficacy of digitally administered intervention by comparing evolution of weight, physical fitness, laboratory measures of metabolic health, blood pressure and other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* obesity with body mass index (BMI) above 30 kg/m^2
* insulin resistance or prediabetes or type 2 diabetes mellitus
* acess to device with internet access (notebook, smartphone, tablet)
* willingness and ability to comply with all scheduled visits, laboratory tests, lifestyle considerations and other study procedures

Exclusion Criteria:

* pregnancy
* steroid treatment
* type 2 diabetes mellitus on insulin therapy
* severe renal and/or hepatic impairment
* any impairments including mental and psychological or conditions which, in the opinion of the investigator, would seriously compromise the integrity of the study
* inability to understand, consent to, or comply with the study protocol for any reason, including inability to read or comprehend Czech language
* inability to comply with study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change in body weight | baseline, three months, six months
  comparison of baseline and end program body weight

SECONDARY OUTCOMES:
change in waist circumference | baseline, three months, six months
  comparison of baseline, three-month and end-program waist circumference between groups
change in body mass index (BMI) | baseline, three months, six months
  comparison of baseline, three-month and end-program body mass index (BMI) between groups
change in haemoglobin A1c | baseline, three months, six months
  comparison of baseline, three-month and end-program haemoglobin A1c values between groups
change in adherence to lifestyle intervention | baseline, three months, six months
  comparison of baseline, three-month and end-program adherence to healthy lifestyle assigned both by subjective (adapted questionnaire) and objective (program usage frequency, attrition) measures between groups
change in blood glucose | baseline, three months, six months
  comparison of baseline, three-month and end-program blood glucose values between groups
change in insulin resistance | baseline, three months, six months
  comparison of baseline, three-month and end-program insulin resistance quantified by HOMA-IR between groups
change in blood pressure | baseline, three months, six months
  comparison of baseline, three-month and end-program blood pressure between groups
change in body composition | baseline, three months, six months
  comparison of baseline, three-month and end-program body composition assessed with the InBody bioelectrical impedance analysis device between groups
change in resting metabolic rate (RMR) | baseline, three months, six months
  comparison of baseline, three-month and end-program resting metabolic rate assessed by indirect calorimetry between groups
change in cardiorespiratory fitness | baseline, three months, six months
  comparison of baseline, three-month and end-program cardiorespiratory fitness assessed by spiroergometry between groups
change in lipid parameters (total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides) | baseline, three months, six months
  comparison of baseline, three-month and end-program levels of total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides between groups
change in fasting insulin levels | baseline, three months, six months
  comparison of baseline, three-month and end-program fasting insulin levels between groups
change in liver function tests | baseline, three months, six months
  comparison of baseline, three-month and end-program standard liver panel (ALT, AST, GGT, ALP) values between groups

OTHER OUTCOMES:
Vitadio usability for HCPs | six months
  The healthcare professionals' (HCPs) user experience from interacting with Vitadio Health, assessed with the User Experience Questionnaire (UEQ)

CONTACTS AND LOCATIONS:
Overall Officials: Katarína Moravcová, MD, Principal Investigator — University Hospital Olomouc
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia